CLINICAL TRIAL: NCT06143202
Title: Feasibility of Continuous Glucose Monitor Use In Hospitalized Youth
Brief Title: Feasibility of CGM Use in Hospitalized Youth
Status: Not yet recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of California, San Francisco (Other); Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 23-1051
Record Dates: First submitted 2023-11-09; First posted 2023-11-22 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Hyperglycemia
Keywords: Hyperglycemia; Continuous glucose monitors; Pediatrics; Hospital; Diabetes
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Pediatric patients with hyperglycemia: Any pediatric patient admitted to the hospital and requiring an endocrine consult for frequent glucose monitoring and hyperglycemia management
  Interventions: Device: Freestyle Libre 3 Continuous Glucose Monitor
- Nursing staff: Nursing staff providing medical care for pediatric patients enrolled in the study.

INTERVENTIONS:
Device: Freestyle Libre 3 Continuous Glucose Monitor — Pediatric participants will wear a blinded Freestyle Libre 3 CGM. Data will not be available, and therefore the device will not be used to modify medical management.
  Groups: Pediatric patients with hyperglycemia

SUMMARY:
This study is assessing the feasibility of a continuous glucose monitor during hospital admissions in youth with hyperglycemia due to diabetes or other underlying conditions that requires frequent glucose monitoring, through pediatric patient/family and nursing staff feedback on their perspectives and usability of the system in the hospital will be assessed through surveys. In addition, retrospective glycemic comparisons between CGM data and POC will be conducted.

DETAILED DESCRIPTION:
Pediatric patients admitted to the hospital for any reason, but require glucose monitoring during the hospitalization will be enrolled in this study. Participant diagnosis can include type 1 diabetes, type 2 diabetes, medication-induced diabetes, cystic fibrosis-related diabetes, or other causes of hyperglycemia that it has been determined by the hospital team requires frequent glucose monitoring, with or without insulin management.

Enrolled participants will wear a blinded continuous glucose monitor for up to 28 days (2 sensors) or until the end of their hospitalization. In addition, enrolled participants will complete a survey to assess their perspectives on the CGM wear experience and interest in future CGM use during hospitalizations. Nursing staff of the enrolled participant will also be invited to complete a survey regarding their perspectives of CGM use in the hospital setting.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be 2 to less than 18 years of age at the time of enrollment.
2. Participants will have a diagnosis of type 1 diabetes, type 2 diabetes, diabetes/hyperglycemia due to an underlying condition (such as in cystic fibrosis, monogenic diabetes), or medication induced diabetes/hyperglycemia (such as steroid-induced hyperglycemia or PEG-asparaginase induced hyperglycemia) and would benefit clinically from close glucose monitoring during hospitalization due to fluctuations in blood glucose values.
3. Participant is expected to be in the hospital for longer than 12 hours after study enrollment with a goal of 36 hours or more as determined by study investigator or trained staff.
4. Participant is willing to wear the continuous glucose monitor for the duration of the hospital admission or the lifespan of a continuous glucose monitor (7-14 days).

Exclusion Criteria:

1. Has had a history of a significant skin reaction to the adhesives of a continuous glucose monitor in the past or concerns that one may occur due to underlying skin conditions (ie severe eczema, uncontrolled psoriasis, etc).
2. Planned MRI or surgery during the study device use (can be enrolled pre or post procedure if sufficient time for sensor wear as determined by investigator [i.e. 24-48 before planned procedure]).
3. Admission to inpatient psychiatry.
4. Pregnancy.
5. Currently using hydroxyurea.
6. A condition that the investigator determines would prevent the patient from participation.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric participants will be admitted to the hospital and have hyperglycemia resulting in an endocrine consult and requiring frequent glucose monitoring.
  Nursing staff providing medical care for the pediatric participant will be invited to complete a survey on usability of the CGM in the hospital setting.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
Retrospective glycemic CGM and point of care comparison | Duration of study, approximately 1 year from study start
  Glycemic data related to time in range, time hypoglycemic, time hyperglycemic and the time of first onset of hypoglycemia and hyperglycemia will be obtained by both CGM and point of care glucose values.

SECONDARY OUTCOMES:
Nursing staff perspectives of CGM use in the hospital | Duration of study, approximately to 1 year from study start
  Surveys will be provided to the nursing staff associated with an enrolled patient participant to obtain qualitative perspectives on the usability of CGMs in the hospital setting
Patient/Family perspectives of CGM use in the hospital | Duration of study, approximately 1 year from study start
  Surveys will be completed by patients/family to evaluate their experience with sensor wear in the hospital, sensor insertion, and goals for glycemic monitoring while in the hospital.
Feasibility of CGM use through assessment of discontinuation and data loss | Duration of study, approximately 1 year from study start
  Identify the frequency and causes of sensor discontinuation as well as information on sensor data loss.
Health economics data | Duration of study, approximately 1 year from study start
  Pilot analysis of health economics data from costs related to glycemic monitoring during the hospitalization.

IPD SHARING:
Plan to Share IPD: No